CLINICAL TRIAL: NCT06018298
Title: Evaluation of Excellence in Italy's Residences for Execution of Security Measures
Brief Title: Evaluation of Excellence in Italy's Residence for Execution of Security Measure
Acronym: ITAL-EE-REMS
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Felice Carabellese, Full Professor of Forensic Psychopathology, University of Bari
Other Study IDs: ITAL-EE-REMS
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Mental Disorder; Recovery; Schizophrenia and Related Disorders; Personality Disorders and Disturbances in Behavior; Personality Disorders, Antisocial; Intellectual Disability, Mild to Moderate
Keywords: Forensic; social dangerousness; therapeutic security
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Personality Disorders; Antisocial Personality Disorder; Intellectual Disability | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapeutic security: assessment of residents in REMS for need for therapeutic security, treatment response relevant to forensic need and forensic recovery.
  Interventions: Other: Treatment as usual (TAU)
- Risk Measures of Need (RISKMON): assessed symptom severity, risk and protective factors for violence, global function, personality factors.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Other: Treatment as usual (TAU) — the components of treatment as usual (TAU) are summarised and assessed by the items of the DUNDRUM-3: physical health, mental health, substance misuse, problem behaviours, self care and activities of daily living, education occupation and creativity, family and intimacy.

SUMMARY:
The model of care for forensic psychiatry in Italy was changed by law (Law 81/2014) so that the six legacy secure forensic hospitals (Judicial Psychiatric Hospitals, OPG) were closed and new secure community residences for the execution of security measures (REMS) were opened in each of the 20 regions of Italy. This transition was in place by 2015. This observational study evaluates the health gains for patients both previously in OPGs and those admitted first to REMS. Health gains assessed include recovery measured by symptoms, function, need for therapeutic security and recovery of legal autonomy.

DETAILED DESCRIPTION:
All those detained in REMS in the twelve month period 2019 to 2020 form the reference population. Samples are assessed for symptom severity (BPRS), global function (GAF), cognitive function (MMSE), risk and protective factors for violence (HCR-20, SAPROF), personality factors (PCL-R), measures of need for therapeutic security (DUNDRUM-1), treatment response relevant to violence and mental illness (DUNDRUM-3) and forensic recovery (DUNDRUM-4).

Outcome measures include violent and challenging behaviour (MOAS), length of stay, conditional (legal) discharge.

ELIGIBILITY:
Inclusion Criteria:

* admitted to REMS
* voluntarily consents to participate

Exclusion Criteria:

* MMSE less than 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents admitted to Residences for the Execution of Security Measures (REMS) under court orders: found by the court to be partially responsible (Penal Code 89) or completely not criminally responsible (Penal Code 88) for a crime and also found socially dangerous (Penal Code 203).
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
length of stay in REMS | date of admission to REMS through study completion, an average of 18 months
  time (days) from admission to move out of REMS
Functional recovery | Date of first, second and third assessments in REMS through study completion, an average of 18 months
  change in GAF over time
violence while in REMS | Date of first, second and third assessments in REMS through study completion, an average of 18 months
  MOAS in the intervals between first, second and third assessments in REMS an average of 18 months
Readmission to REMS | date of discharge from REMS to date of readmission to REMS, if any.
  time (days) until readmission to REMS following discharge from REMS an average of 18 months

SECONDARY OUTCOMES:
conditional discharge | date of assessment to date of conditional discharge an average of 18 months
  time (days) from date of assessment to date of conditional discharge

OTHER OUTCOMES:
Death | from date of admission to date of death while in REMS, if any up to two years
  death while in REMS, if any

CONTACTS AND LOCATIONS:
Overall Officials: Felice F Carabellese, MD, Study Director — University of Bari; Lia Parente, PsyD, Principal Investigator — University of Bari; Harry G Kennedy, MD, Principal Investigator — University of Dublin Trinity College (TCD); Mary Davoren, MD, Principal Investigator — University of Dublin Trinity College (TCD)
Locations (1):
- University of Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
In view of the sensitive nature of the data, aggregated anonymised data may be provided to accredited researchers on a case by case basis.

REFERENCES:
- [Background] Carabellese F, Parente L, Kennedy HG. Reform of Forensic Mental Health Services in Italy: Stigma and Blaming the Messenger: Hermenoia. Int J Offender Ther Comp Criminol. 2024 Nov;68(15):1505-1524. doi: 10.1177/0306624X221113531. Epub 2022 Jul 21. PMID 35861358
- [Background] Flynn G, O'Neill C, McInerney C, Kennedy HG. The DUNDRUM-1 structured professional judgment for triage to appropriate levels of therapeutic security: retrospective-cohort validation study. BMC Psychiatry. 2011 Mar 16;11:43. doi: 10.1186/1471-244X-11-43. PMID 21410967
- [Background] Jeandarme I, Habets P, Kennedy H. Structured versus unstructured judgment: DUNDRUM-1 compared to court decisions. Int J Law Psychiatry. 2019 May-Jun;64:205-210. doi: 10.1016/j.ijlp.2019.04.006. Epub 2019 May 1. PMID 31122631
- [Background] KENNEDY, H. G. 2002. Therapeutic uses of security: mapping forensic mental health services by stratifying risk. Advances in Psychiatric Treatment, 8, 433-443.DOI: https://doi.org/10.1192/apt.8.6.433
- [Background] O'Neill C, Smith D, Caddow M, Duffy F, Hickey P, Fitzpatrick M, Caddow F, Cronin T, Joynt M, Azvee Z, Gallagher B, Kehoe C, Maddock C, O'Keeffe B, Brennan L, Davoren M, Owens E, Mullaney R, Keevans L, Maher R, Kennedy HG. STRESS-testing clinical activity and outcomes for a combined prison in-reach and court liaison service: a 3-year observational study of 6177 consecutive male remands. Int J Ment Health Syst. 2016 Oct 11;10:67. doi: 10.1186/s13033-016-0097-z. eCollection 2016. PMID 27766115
- [Background] Williams HK, Senanayke M, Ross CC, Bates R, Davoren M. Security needs among patients referred for high secure care in Broadmoor Hospital England. BJPsych Open. 2020 Jun 2;6(4):e55. doi: 10.1192/bjo.2020.35. PMID 32482202
- [Background] Carabellese F, Felthous AR. Closing Italian Forensic Psychiatry Hospitals in Favor of Treating Insanity Acquittees in the Community. Behav Sci Law. 2016 Mar;34(2-3):444-59. doi: 10.1002/bsl.2234. PMID 27256003
- [Background] Catanesi R, Mandarelli G, Ferracuti S, Valerio A, Carabellese F (2019). The new Italian residential forensic psychiatric system (REMS). A one-year population study. Italian Journal of Criminology - Special Number, Vol.13.
- [Background] Cura e controllo. Come cambia la pericolosità sociale psichiatrica R Catanesi, FF Carabellese, I Grattagliano - Giornale Italiano di Psicopatologia, 2009
- [Background] Carabellese F, Felthous AR, Rossetto I, La Tegola D, Franconi F, Catanesi R. Female Residents with Psychopathy in a High-Security Italian Hospital. J Am Acad Psychiatry Law. 2018 Jun;46(2):171-178. doi: 10.29158/JAAPL.003744-18. PMID 30026395
- [Background] Comportamento violento in una coorte di pazienti psichiatrici: rischio psicosociale e fattori protettivi F Carabellese, C Candelli, D La Tegola, R Buzzerio… - Rassegna italiana di criminologia, 2015
- [Background] Gualtieri G, Traverso S, Pozza A, Ferretti F, Carabellese F, Gusinu R, Coluccia A. Clinical risk management in High-Security Forensic Psychiatry Residences. Protecting patients and health professionals: perspectives and critical issues of the Law 81/2014. Clin Ter. 2020 Mar-Apr;171(2):e97-e100. doi: 10.7417/CT.2020.2196. PMID 32141478
- [Background] OPG di chiusura: strumenti diagnostici per criminali malati di mente socialmente pericolosi. Dalla valutazione medico-psichiatrica al trattamento F Carabellese - Rassegna Italiana di Criminologia, 2017
- [Background] Assessing the needs of patients in secure settings: a multi-disciplinary approach P Pierzchniak, F Farnham, N Taranto, D Bull, H Gill… - The Journal of Forensic Psychiatry, 1999
- [Background] Models of care in forensic psychiatry HG Kennedy - BJPsych Advances, 2022
- [Derived] Parente L, Carabellese F, Felthous A, La Tegola D, Davoren M, Kennedy HG, Carabellese FF. Italian Evaluation and Excellence in REMS (ITAL-EE-REMS): appropriate placement of forensic patients in REMS forensic facilities. Int J Ment Health Syst. 2024 Nov 2;18(1):33. doi: 10.1186/s13033-024-00647-5. PMID 39488677